CLINICAL TRIAL: NCT07366606
Title: Development of a Thromboelastography-Based Algorithm for Targeted Bleeding Management in Open Heart Surgery: An In Vitro Clinical Study
Brief Title: Bleeding Management İn Open Heart Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Serkan Uckun (Other)
Responsible Party: Sponsor-Investigator, Serkan Uckun, assistant professor, Balikesir University
Organization: Balikesir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AHTEG
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Thromboelastography (TEG); Open Heart Surgery; Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The decision regarding blood and blood product transfusions will be made based on clinical observation by an anesthesiologist, which is our current routine practice.
- Group T (Active Comparator): Blood clotting tests are performed with the device.
  Interventions: Diagnostic Test: Blood Product

INTERVENTIONS:
Diagnostic Test: Blood Product — R time, the time from the start of the test until the graph width reaches 2 mm (5-10 minutes), reflects the activity of clotting factors.
  K time, the time from the end of R until the width reaches 20 mm (1-3 minutes), represents the clot formation time and rate.
  alpha angle (53-72 degrees) represents fibrinogen function, maximum amplitude is related to platelet function (50-70 mm), represents maximum clot strength.
  lysis rate -30 (0% -8%) represents the clot lysis rate 30 minutes after MA, indicating whether hyperfibrinolysis is present.
  Arms: Group T

SUMMARY:
This study aims to develop an algorithm that can guide targeted bleeding management through thromboelastography (TEG) viscoelastic testing performed on blood samples from patients undergoing open heart surgery. The goal is to develop an algorithm that supports targeted bleeding management based on TEG parameters. The study is prospective, in vitro, and non-invasive. The material will consist of residual blood samples from open heart surgery patients. Analyses will be performed using TEG parameters (R time, K time, MA, LY30). Patients will be randomized using a closed-envelope method and divided into two groups: anesthesiologist standard clinical observation-control (Group K) and anesthesiologist standard clinical observation and TEG analysis (Group T). The sample size is 70 patients per group. From an ethical standpoint, this study uses anonymous data without additional blood collection and ensures patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo open heart surgery
* Patients who have given informed consent

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients with known congenital coagulation disorders
* Patients with a known history of bleeding diathesis
* Patients receiving uninterrupted anticoagulant therapy at an optimal time
* Patients with renal failure under dialysis treatment
* Patients with active malignancy
* Patients who did not provide informed consent

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Targeted coagulation therapy | A total of three measurements will be take After induction of anesthesia (Between 15 and 30 minutes of the operation) During cardiopulmonary bypass (2 hours after the start of surgery) Following cardiopulmonary bypass (4 hours after the start of surgery)
  Measurement of R time using thromboelastography Measurement of K time using thromboelastography Measurement of maximum amplitude using thromboelastography

SECONDARY OUTCOMES:
Use of blood products | Anesthesia continues during cardiopulmonary bypass exit (4 to 5 hours after surgery)
  Optimizing the use of fibrinogen, platelets, and fresh frozen plasma by combining thromboelastography measurements with clinical interpretation